| Official Title | A Phase Ib Open-label Study Evaluating the Safety and |
|---|---|
| | Efficacy of NKTR-255 in Combination with |
| | CD19-Directed CAR-T Cell Therapy in Patients with |
| | Relapsed/Refractory (R/R) Large B-Cell Lymphoma (LBCL) |
| NCT Number | NCT05359211 |
| Document Type | Informed Consent Form |
| <b>Document Date</b> | 9/28/2024 |

# FRED HUTCHINSON CANCER CENTER UNIVERSITY OF WASHINGTON SCHOOL OF MEDICINE

A Phase Ib Open-label Study Evaluating the Safety and Efficacy of NKTR-255 in Combination with CD19-Directed CAR-T Cell Therapy in Patients with Relapsed/Refractory (R/R) Large B-Cell Lymphoma (LBCL)

| Sponsor-Investigator | Professional Title | Phone Number |
|---------------------------|---------------------------------|----------------|
| Alexandre V. Hirayama, MD | Assistant Professor, Fred Hutch | 206-667-6909 |
| | Assistant Professor, UW | |
| Investigators | | |
| Jordan Gauthier, MD | Associate Professor, Fred Hutch | 206-667-2713 |
| | Associate Professor, UW | |
| Biostatistician | | |
| Qian "Vicky" Wu, PhD | Assistant Professor, Fred Hutch | 206-667-3358 |
| Research Staff | | |
| Mike L. Miller | Clinical Research Coordinator | (206) 667-7782 |
| Allie Sullivan, RN | Research Nurse | (206) 667-5979 |

**EMERGENCY (24-HOUR) PHONE: 206-598-8902** 

If you are serving as a legally authorized representative or a guardian, the terms "participant", "you", and "your" refer to the person for whom you are providing consent for.

## Important things to know about this study.

You are invited to participate in a research study. The purpose of this research is to find out if NKTR-255 (a drug that can promote inflammatory and protective immune responses in your body) can help promote the survival and effects of chimeric antigen receptor (CAR)-T cell therapy.

The study is conducted by Fred Hutch researchers, who are the Sponsor-Investigator/s of the study. Nektar Therapeutics, a biopharmaceutical company, has created and will provide the study drug, NKTR-255, and financially supports this study; but is not the regulatory sponsor of the study.

NKTR-255 is an investigational treatment meaning it has not yet been approved for sale or use to the public by the United States Food and Drug Administration.

If you agree to join the study, you will receive up to 3 intravenous (IV) infusions of NKTR-255, over the course of 9 weeks, starting approximately 10 or 14 days after you receive lisocabtagene maraleucel (lisocel; Breyanzi®) infusion for your cancer. Which study cohort and/or dose level you participate in on the study, will be determined by your Study doctor and depends on the timing in which you enroll in the study. The study doctor will confirm which cohort and dose level of NKTR-255 you will participate on once you are determined to be eligible for the study. The frequency and number of NKTR-255 infusions you receive may also be adjusted based on how you are responding to the treatment and at the discretion of the researchers completing this study.

You would remain in this study for approximately 1 year to complete short term follow-up. If you decide to leave the study early, you will be asked to complete an end of treatment visit (EOT). You may complete long-term follow-up per standard of care as required for your liso-cel treatment. This will be discussed with you by your treating physician.

We do not know if NKTR-255 will help to treat your cancer or enhance your CAR-T cell therapy. NKTR-255 may cause side effects such as fever, chills, nausea, headache, fatigue (tiredness). Liso-cel could also cause side effects such as severe fever, nausea, headache, and temporary changes in behavior (known as neurologic toxicities). Other possible side effects are described below in this form.

You do not have to join this study. You could choose not to participate in the study and just receive CAR-T cell therapy per standard of care. If you choose not to participate in this study, it will not affect your routine medical care or your standard of care CAR-T cell therapy.

We will give you details about the purposes, procedures, risks, and possible benefits related to this study. We will explain other choices that you have. We will also give you any other information that you need in order to make an informed decision about joining this study.

Following is a more complete description of this study. Please read this description carefully. Afterwards, you can ask questions that will help you decide whether to join the study. If you join this study, we will give you a signed copy of this form to keep for future reference.

## We invite you to join this research study.

We invite you to join this research study because you have large B-cell lymphoma (LBCL) that has either recurred or not responded to conventional chemotherapy or other treatments, and you are about to get treatment with lisocabtagene maraleucel (liso-cel; Breyanzi®), a CAR-T cell therapy.

Research is not the same as treatment or medical care. The purpose of a research study is to answer scientific questions. We will enroll up to 24 people with LBCL for this research study.

You do not have to be in this study. You are free to say "yes" or "no", and you are also allowed to change your mind after joining. There is no penalty or loss of benefits if you say no. Whatever you decide, your regular medical care will not change.

# Why are we doing this study?

We are doing this study to see if a drug called NKTR-255, a cytokine (which is a type of protein your body naturally makes) could improve your CAR-T cell therapy. Specifically, it is a type of cytokine called Interleukin-15 (IL-15) that can help with protective immune responses and help fight diseases. IL-15 may help with the growth, survival, and efficacy of CAR-T cells, like liso-cel.

This study is investigating the safety and tolerability of NKTR-255 in combination with liso-cel immunotherapy in treating your disease. This study is also looking to find out the optimal starting day to give NKTR-255 to patients. The study doctor will explain to you in more detail which study day you may receive.

# What research tests, procedures, and treatments are done in this study?

If you decide to join this study, we will do the following research tests and procedures, which may be performed in addition to your usual care. Where possible we will try to schedule the times and locations of research tests at the same time as the tests done as part of your usual care.

To determine if you are eligible for this study, a number of routine tests will be evaluated. This will include routine blood tests, including testing for blood grouping, viruses like hepatitis and HIV, complete blood counts, pregnancy test (if applicable), and metabolic function panels. You will have medical tests done to evaluate your heart, lungs, and other organs (if necessary). If any of these tests have to be repeated as part of the study, they will be considered outside of your standard of care.

There are several parts to this study. Some of the procedures completed will be part of your standard of care for liso-cel. Other assessments will be considered research only as part of your NKTR-255 infusion, which is the investigational treatment on this study.

- 1) Screening/Pretreatment
- 2) Liso-cel infusion and evaluations
- 3) NKTR-255 infusion(s) and evaluations
- 4) NKTR-255 post-infusion evaluations
- 5) Follow-up evaluations

#### **Screening/Pretreatment**

You will complete the evaluations below as part of your standard of care for liso-cel treatment. Results of tests and procedures conducted as your standard of care may be used for this study. However, if any of the following tests or procedures are completed more than 28 days prior to your leukapheresis, you may need to have them repeated for research purposes:

- Medical history and physical examination, including height and weight.
- Review of your ability to perform everyday tasks.
- If you are female of childbearing potential, you will have a blood pregnancy test done.
- Routine laboratory blood tests.

Where possible, some of the below evaluations will be completed per standard of care. Due to clinical or logistical factors, it is possible to have variations in completion of standard of care evaluations. The following events should be conducted:

- Leukapheresis: In order to receive your liso-cel product, you will undergo a leukapheresis procedure. Your treating physician will discuss this with you in more detail including any risks associated with this procedure. Approximately 5 mL of your leukapheresis product may be collected for this study for research purposes.
- **Tumor Biopsy:** A tumor biopsy may be obtained. There are two reasons you may undergo a tumor biopsy:
  - o **Clinical biopsy:** A tumor biopsy may be necessary for your clinical care; if obtained, a research sample may be sent to the research lab.
  - Research tumor biopsies: If you have a tumor that your doctor thinks can be safely biopsied, we would like to perform a biopsy procedure to get some tumor tissue for research. Similarly, should your doctor determine that a biopsy cannot be performed safely for clinical reasons, biopsies may be cancelled or rescheduled. Your doctor will explain the process and risks to you and tell you which tumor they feel is best to biopsy. We would like to collect research biopsies during 1) pre-treatment prior to receiving your chemotherapy and liso-cel infusion; 2) within 4 weeks after you receive your liso-cel infusion 3) within 4 weeks after your first NKTR-255 infusion; and 4) in the event of a persistent mass, or your disease progresses. You will be asked to provide consent to these optional biopsies at the end of this form.
- The study team may also request some archival tissue from a previously collected biopsy for research if available.
- Imaging studies: You may have CT (Computed Tomography) scans with or without PET (Positron Emission Tomography) scans to determine the amount of disease you have prior to starting chemotherapy. This may be omitted if you have already had imaging completed within 30 days of your scheduled liso-cel infusion.
- **Blood tests:** You may have up to 45 mL (approximately 3 tablespoons) of blood collected for research purposes for this study. Some of the samples will be stored for analysis later or for future research.
- Other routine medical tests will be done to evaluate your heart, lungs, and other organs to make sure it is safe for you to participate in the study. These may include a physical exam, neurological

exam, electrocardiogram (ECG), echocardiogram (ECHO) or a multi-gated acquisition (MUGA), pregnancy test if applicable and laboratory blood tests.

- A lumbar puncture (spinal tap) for cerebrospinal fluid (CSF) may be collected if clinically indicated.
- If you have any other tissue collected, a portion may be requested for this research study.

#### Liso-cel infusion and evaluations

The following evaluations should be done on the day you receive your liso-cel infusion as part of routine clinical evaluations:

- Medical history and physical examination.
- Review of your ability to perform everyday tasks.
- Routine laboratory blood tests.
- You will have your vital signs monitored which includes oxygen saturation, blood pressure, and heart rate before, during, and after the infusion.

The following evaluations will be done for purposes of this research study:

- **Blood tests:** You may have up to 45 mL (approximately 3 tablespoons) of blood collected for research purposes for this study. Some of the samples will be stored for analysis later or for future research.
- **Liso-cel infusion product:** After you receive your liso-cel infusion we may request to collect any leftover product that remains in the infusion bag or tubing for this research study.

#### **Evaluations after liso-cel infusion**

After liso-cel infusion, you may have the following tests and procedures. If you are unable to receive your NKTR-255 infusion, you will still have the following evaluations done.

- History and physical examination (with a neurological exam if clinically indicated) 1 day after the liso-cel infusion and at least weekly until you receive your first NKTR-255 infusion.
- Review of your ability to perform everyday tasks.
- Routine laboratory blood tests.
- **Blood tests:** On days 1, 3, 7, 10, and 14, you may have up to 45 mL (approximately 3 tablespoons) of blood collected for research purposes for this study. Some of the samples will be stored for analysis later or for future research.
  - o If you experience any signs of toxicity symptoms from your liso-cel infusion, additional blood samples may be collected in-between the previously indicated time points. Depending on how you are feeling, it is possible that at multiple time points you may have an additional 45 mL (approximately 3 tablespoons) of blood collected.
- A lumbar puncture (spinal tap) for cerebrospinal fluid (CSF) may be collected if clinically indicated.
- If you have any other tissue collected for clinical purposes, a portion may be requested for this research study.

- If available, your leftover liso-cel product may be collected from the product container bag after your infusion is complete.
- If you consent to having additional, optional tumor biopsies collected, you may have a tumor biopsy performed at this time (within 4 weeks of your liso-cel infusion). Timing will be discussed with you by the study doctor.

#### **Evaluations on the day of each NKTR-255 infusion**

You will receive your first NKTR-255 infusion on either day 10 or 14 after your liso-cel treatment. You will receive NKTR-255 approximately every 3 weeks via intravenous (IV) infusion. You may receive up to 3 infusions of the study product. The following will occur on the day of each NKTR-255 infusion.

- History and physical examination including weight (with neurological exam if clinically indicated).
- Review of your ability to perform everyday tasks, review of your current medications and how well you are feeling.
- Routine laboratory blood tests.
- ECG.
- **Blood tests:** Before, during and after your first NKTR-255 infusion you will have blood samples collected. Approximately 63 mL (approximately 5 tablespoons) of blood will be collected for research purposes for this study. Some of the samples will be stored for analysis later or for future research. If it is not your first NKTR-255 infusion, you may have slightly less blood obtained, approximately 50-55 mL (approximately 4.5 tablespoons).
- You will have your vital signs monitored which includes oxygen saturation, blood pressure, and heart rate before, during, and after the infusion.

#### NKTR-255 Cycles 1 and 2 post-infusion evaluations

After each NKTR-255 infusion for cycle 1 and cycle 2, you will need to complete some post-infusion evaluations. After your first and second infusion of the NKTR-255 study product you will follow the below post-infusion evaluations schedule:

- History and physical examination on the day after your infusion day, twice weekly for the first 2
  weeks after NKTR-255 infusion, then at least weekly. You may also have a neurological exam
  performed.
- Review of your ability to perform everyday tasks, review of your current medications and how well you are feeling.
- Routine laboratory blood tests completed twice weekly for the first 2 weeks after NKTR-255 infusion and then at least weekly.
- **Blood tests:** On days 1, 3, 7, 10, and 14 after NKTR-255 infusion, you may have up to approximately 55 mL (approximately 4.5 tablespoons) of blood collected for research purposes for this study on each visit day. Some of the samples will be stored for analysis later or for future research.
  - If you experience any signs of toxicity symptoms from your liso-cel infusion, additional blood samples may be collected in-between the previously indicated time points. Depending on how you are feeling, it is possible that at multiple time points

you may have an additional 48 mL (approximately 3 tablespoons) of blood collected over multiple time points.

- If you consent to having additional, optional tumor biopsies collected, you may have a tumor biopsy performed at this time (within 4 weeks of your first NKTR-255 infusion). Timing will be discussed with you by the study doctor.
- If you have any other tissue collected for clinical purposes, a portion may be requested for this research study.

For the purposes of restaging your disease, the following may be done as part of your standard of care after liso-cel treatment:

- CT and PET scans.
- A bone marrow aspirate and biopsy may be collected if clinically indicated.
- A lumbar puncture (spinal tap) for cerebrospinal fluid (CSF) may be collected if clinically indicated.

If you are able to receive your third infusion of NKTR-255 study product, you will follow the below post-infusion evaluations schedule after each infusion:

- History and physical examination at least weekly after NKTR-255 infusion. You may also have a neurological exam performed.
- Review of your ability to perform everyday tasks, review of your current medications and how well you are feeling.
- Routine laboratory blood tests completed at least weekly for the first 3 weeks after NKTR-255 infusion.
- **Blood tests:** will be collected approximately weekly for up to 3 weeks after NKTR-255 infusion. You may have up to 45 mL (approximately 4 tablespoons) of blood collected for research purposes for this study. Some of the samples will be stored for analysis later or for future research.
  - O If you experience any signs of toxicity symptoms from your liso-cel infusion, additional blood samples may be collected in-between the previously indicated time points. Depending on how you are feeling, it is possible that at multiple time points you may have an additional 45 mL (approximately 3 tablespoons) of blood collected.
- If you consent to having additional, optional tumor biopsies collected, you may have a tumor biopsy performed at this time in case of persistent mass, progression, or relapse. Timing will be discussed with you by the study doctor.
- If you have any other tissue or fluids collected for clinical purposes a portion may be requested for this research study.

For the purposes of restaging your disease, the following may be done as part of your standard of care after liso-cel treatment:

• CT and PET scans at approximately every 3 months.

#### **Follow-up evaluations**

The following evaluations will occur approximately 30 days after you receive your last infusion of NKTR-255 or as part of an end of treatment (EOT) visit and then approximately at 3, 6, 9, and 12 months after liso-cel infusion:

- Physical examination (with neurological exam if clinically indicated).
- Blood draw for routine laboratory tests.
- **Blood tests:** approximately 3 months after the last NKTR-255 dose and on months 3, 6, 9, and 12 after liso-cel infusion, you may have up to 52 mL (approximately 4 tablespoons) of blood collected for research purposes for this study. Some of the samples will be stored for analysis later or for future research.
  - o If you experience any signs of toxicity symptoms from your liso-cel infusion, additional blood samples may be collected in-between the previously indicated time points. Depending on how you are feeling, it is possible that at multiple time points you may have an additional 48 mL (approximately 3 tablespoons) of blood collected.
- If you consent to having additional, optional tumor biopsies collected, you may have a tumor biopsy performed at this time in case of persistent mass, progression, or relapse. Timing will be discussed with you by the study doctor.
- If you have any other tissue collected for clinical purposes a portion may be requested for this
  research study

For the purposes of restaging your disease, the following may be done as part of your standard of care after liso-cel treatment:

• CT and PET scans at approximately 3, 6, 9, and 12 months after your liso-cel infusion as clinically indicated.

# Long term Follow-up

After you complete your 12-month visit or an end of treatment (EOT) visit, you will have completed the main treatment study. You will be followed for long-term follow-up per institutional standard of care for your liso-cel infusion. You may be contacted annually for up to 15 years. You may have to sign an additional consent for this and your clinical physician will discuss this with you.

# How long would you stay in this study?

You will be actively participating in the study for approximately one year from the day of liso-cel infusion. We will also follow the results of restaging that will be performed by your treating oncologist.

The study doctor or your doctor may take you out of this study at any time, whether you want to leave the study or not. This would happen if:

• They think it is not in your best interest to continue in the study.

- You are not able or willing to follow study procedures.
- The whole study is stopped.

If you are thinking about dropping out of this study, please tell the study doctor. The doctor can tell you about the effects of stopping.

If you withdraw from the study for any reason, you will be asked to complete an end of treatment visit (EOT) within 7 days of informing us you would like to stop the study. Previously collected information would remain in the study records and would be included in the analysis of results. This information could not be removed from the study records.

### What are the side effects (risks)?

In this part of the consent form, we describe the side effects we expect from NKTR-255 and from the tests in this study.

With any new treatment or combination of treatments, there may be side effects that we do not know about and cannot predict. NKTR-255 is an investigational product that has been used in research trials before. This study will be the first time NKTR-255 is given in combination with a CAR-T cell therapy (liso-cel).

The side effects associated with NKTR-255 are listed below. We do not know if combining NKTR-255 with liso-cel will change these side effects. Combining NKTR-255 with liso-cel could worsen side effects of either product or have other effects that we do not know about.

If we learn about any new side effects, we will tell you. We carefully watch everyone in the study for side effects. If you want more information about side effects and risks, ask the doctor or nurse.

You should talk to your doctor about any side effects that you have while you are in this study.

If they occur, side effects may be mild or very serious. Your health care team may give you medicines to help lessen side effects.

#### Risks of NKTR-255

Below are risks associated with NKTR-255 as experienced in other research studies:

- Flu-like symptoms (may include symptoms of fever and chills)
- Fatigue (tiredness)
- Rash
- Itching skin
- Low blood pressure
- Facial swelling or swelling of the area beneath the skin (may include hives, swelling of eye, lip, mouth, and tongue)
- Muscle or joint pain
- Fainting (may occur due to low blood pressure)
- Cytokine-related toxicities: symptoms may include flu-like symptoms, fevers, chills, rash, itchy
  skin, fatigue, low blood pressure, joint pain, muscle pain, abnormal kidney function tests, and
  abnormal liver enzyme tests.
- Infusion-related reaction or allergic reaction (discussed in more detail below)
- Cytokine release syndrome (discussed in more detail below)

• Immune effector cell-associated neurotoxicity syndrome (ICANS -discussed in more detail below)

#### Your study doctor will also watch you closely for the following potential side effects:

- Cytokine Release Syndrome (CRS): When modified T cells grow in your body and attack cancer cells, they release inflammatory chemicals called cytokines. The release of large amounts of these cytokines can lead to fever, nausea, headache, fast heart rate, changes in blood pressure, shortness of breath, and low oxygen levels in the blood/body. If you are not in the hospital and develop a fever, you should call your study doctor immediately.
- Immune effector cell-Associated Neurotoxicity Syndrome (ICANS) ICANS is a recognized consequence of immune-effector cell therapy. On this study, the potential exists for ICANS when NKTR-255 is administered following CAR-T cell therapy (such as liso-cel). ICANS may include, but is not limited to, symptoms such as encephalopathy (brain swelling), difficulty with paying attention, speech (finding the right words to say) or handwriting, confusion, agitation, sleepiness, seizures, motor weakness, and tremors. ICANS is usually reversible but can be irreversible or fatal.
- Eosinophilic disorder (disorders associated with elevated eosinophil count in blood, a type of white blood cell): your study doctor will closely monitor your blood counts while you are receiving NKTR-255. If you have a high eosinophil count, your doctor may ask you if you have experienced the following symptoms, including but not limited to: rash, wheezing/difficulty breathing, abdominal pain, chest pain, ankle swelling, and confusion.
- Reactions associated with infusion (events occurring during or within 24 hours of infusion): symptoms may include fever, chills, shortness of breath, low blood pressure, headache, facial swelling, rash, itchy skin, muscle pain and joint pain and other allergic-like reactions.
- Neutropenia (abnormal count of a type of white blood cells, called neutrophils): your doctor will closely monitor your blood counts while you are receiving NKTR-255.
- Thrombocytopenia: is a condition in which you have a low blood platelet count. Platelets are colorless blood cells that help in blood clotting. Symptoms and signs of thrombocytopenia are easy or excessive bruising, increased bleeding time and fatigue.
- Infections: can occur if you have a low number of lymphocytes and neutrophils in the blood. Lymphocytes and neutrophils are the white blood cells of the immune system that are involved in protecting your body from infections. Infections may be caused by bacteria or virus including reactivation of previous viral diseases. You should immediately let your study doctor know if you start experiencing any of the following symptoms: fever, chills, feeling tired or fatigued, headache, nausea, vomiting, shortness of breath, pain, confusion, etc.
- QT/QTc prolongation: a longer than usual measurement of one electrical property of your heart. Symptoms may be dizziness, lightheadedness, heart palpitations, fast heartbeat, and shortness of breath.

- Allergic Reactions to NKTR-255: You may have an allergic reaction to NKTR-255, such as itching; skin rash; facial swelling; swelling inside the throat with difficulty breathing; and an acute or sudden drop in blood pressure. The sudden drop in blood pressure may lead to shock with loss of consciousness and/or possible seizures, including the possibility of death. If any of the above symptoms of an allergic reaction occurs, seek medical attention immediately.
- Other Reactions: You may also experience dizziness and nausea. Other rare or unknown side effects to study drug could possibly occur, including life threatening reactions.

#### Risks of other study procedures

Where possible, we will schedule study blood tests to take place at the same times as your regular clinical tests to minimize any risks and discomfort. If you have the tests done separately, the extra risks are as follows.

#### **Blood tests**

The risks of blood tests depend on whether the blood is taken by needle directly from a vein or from a device, such as a Port or Hickman catheter, that stays in place for blood tests. If blood is taken from a Hickman catheter, there is usually no pain or bruising.

Likely side effects ( $\geq 20\%$ ) of blood tests are:

- Temporary discomfort if blood is taken straight from a vein.
- A small bruise or redness at the site from which the blood was taken.

Less likely side effects (3-20%) of blood tests are:

- Fainting, sweating, or feeling sick in the stomach that gets better when you lie down and rest.
- Bruising larger than a "quarter" coin.

Rare but serious side effects (< 3%) of blood tests are:

- Infection from the blood draw.
- Injury to blood vessels, nerves, or other structures near the blood draw site.

#### **CT/PET Scans**

Some of the tests that you will have in this research study will expose you to radiation. Everyone receives a small amount of radiation every day called "background radiation". This radiation is natural and comes from space, air, water, soil, and the food you eat. Each year you are exposed to about 3 milliSieverts (mSv) of this background radiation. A milliSievert is a unit of radiation dose. For comparison, the estimated radiation dose from each of these tests is listed below.

• PET/CT: 19 mSv

#### **Tumor Biopsy**

Likely side effects ( $\geq 20\%$ ) of tumor biopsy procedures are:

- · Bruising.
- Pain or discomfort from where the needle punctures the skin.

Less likely side effects (3-20%) of tumor biopsy procedures are:

- Infection from the biopsy.
- Injury to blood vessels, nerves, or other structures.

Rare but serious side effects (< 3%) of tumor biopsy procedures are:

• Serious reaction to the anesthesia drugs.

#### Reproductive risks

NKTR-255 may involve unknown risks to an embryo, fetus (unborn baby) or nursing infant. Therefore, you could not join this study if you are pregnant, if you are planning to become pregnant, or if you are breast-feeding.

If you join this study, you would have to use an effective method of birth control from the time this form is signed until at least 1 month after the last dose of NKTR-255. If you are already using a method of birth control, you would have to check with the study doctor or a member of the study staff to make sure it is acceptable.

If you became pregnant after joining this study, you would have to notify the study doctor immediately.

The effects of NKTR-255 on fathering a child are also unknown. Men who join this study must also agree to use one or more forms of effective and acceptable birth control from the time this form is signed until at least 1 month after the last dose of NKTR-255.

#### What are the benefits?

We hope that combining NKTR-255 with your liso-cel treatment will help with how well liso-cel works in treating your cancer, however, at this time we do not know if it will. Combining NKTR-255 with liso-cel treatment is investigational. We hope the information from this study will help us find out if NKTR-255 can help patients who receive CAR-T cells in the future.

# You have other choices besides this study.

You do not have to join this study. You are free to say "yes" or "no". Your regular medical care would not change if you say "no".

If you do not join this study, you have other choices for treatment. Each of these choices has risks and benefits. Talk to your doctor about your choices.

Your other choices may include:

- Treatment with liso-cel only, not as part of this research study.
- Supportive care.
- A different research study.
- Enrollment in this study may exclude you from other research studies.

## Protecting Privacy as an Individual and the Confidentiality of Personal Information

If you join this study, some people or organizations might need to look at your medical records and research records for quality assurance or data analysis. They include:

- Researchers involved with this study.
- Institutional Review Boards (IRB), including the Fred Hutchinson Cancer Center IRB. An IRB is a group that reviews the study to protect your rights as a research participant.
- Fred Hutchinson Cancer Center, University of Washington.
- Office for Human Research Protections, Food and Drug Administration, and other agencies as legally required.
- Nektar Therapeutics, a biopharmaceutical company providing the study drug, NKTR-255 and financial support for this study, and any of their agents or collaborators.

We will do our best to keep your personal information confidential. But we cannot guarantee total confidentiality. Your personal information may be given out if required by law. For example, workplace safety rules may require health workers to contact you about lab tests. Or a court may order study information to be disclosed. Such cases are rare.

We will not use your personal information in any reports about this study, such as journal articles or presentations at scientific meetings.

Policies of the University of Washington (UW Medicine) and the Fred Hutchinson Cancer Center (FHCC) require that certain information about participation in this research must be included in permanent medical records.

If you join this study but do not already have a medical record at UW Medicine or FHCC, we would create a record even if the only connection with UW Medicine or FHCC involves this research study.

The information in the permanent medical record would include:

- Name of the study.
- Name of the group or company that is paying for the research.
- The number the group or company assigned to this study.
- The name of the researcher.
- The name of the study coordinator.
- Contact phone number for the study.

- Contact email address for the study.
- Emergency phone number for the study.
- A copy of this consent form.

If you join this study, information about your participation would be made part of your permanent medical record. This information would include a copy of this consent form. If you authorize others to see your medical record, they would see a copy of this consent form.

## How is my genetic information protected?

A federal law called the Genetic Information Nondiscrimination Act (GINA) helps protect genetic information about people who join research studies.

GINA restricts access to genetic information so that it cannot be used for health insurance coverage decisions. GINA prevent health insurance companies or group health plans from

- Asking for genetic information obtained in research studies, or
- Using genetic information when making decisions regarding your eligibility or premiums.

GINA *does not* help or protect against genetic discrimination by companies that sell life, disability or long-term care insurance.

## Would we pay you if you join this study?

You and/or your caregiver are eligible for reimbursement of up to \$6000 for travel expenses (i.e. airfare, mileage, parking, overnight accommodations and food) related to your participation in this study from the time of your consent to 30 days post your final NKTR-255 infusion. You will need to give us receipts that clearly show your costs.

It is possible that through the use of your samples collected in this study a commercial product may be developed. Nektar Therapeutics, Fred Hutchinson Cancer Center, other researchers, or companies may patent or sell discoveries that result from this research. Neither Nektar Therapeutics, study doctor, nor study site will compensate you if this occurs.

# Would you have extra costs if you join this study

If you join this study, you would have some extra costs. You or your insurer will have to pay for the routine costs of treating your cancer in this study including your liso-cel treatment. Check with your insurer before you join this study as some insurers will not pay for research. Taking part in the study may lead to extra costs for you or your insurance company because of the possibility of additional hospitalizations, procedures, and blood tests.

The NKTR-255 you receive during this study will be provided to you at no cost by Nektar Therapeutics.

If you have any questions concerning your costs, financial responsibilities, and or medical insurance coverage for this activity, please ask your physician or contact the Patient Financial Services Department at (206) 606-6226.

# What if you get sick or hurt after you join this study?

For a life-threatening problem, call 911 right away or seek help immediately. Contact your study doctor when the medical emergency is over or as soon as you can.

For all other medical problems or illness related to this research, immediately contact the Immunotherapy clinic by calling (206) 606-6000. They will treat you or refer you for treatment. You or your health insurance may have to pay for the treatment. Nektar Therapeutics will pay for the reasonable costs of medical care for an injury or illness caused by a defect in the manufacture or design of the study drug, NKTR-255.

You or your insurer will be billed for treatment of problems or complications that result from your condition or from standard clinical care.

You would not lose any legal right to seek payment for treatment if you sign this form.

## What will my information and/or tissue samples be used for?

Your information and blood or tissue samples will be used for the purposes of this study.

Your blood and tissue samples might help researchers develop new products. This research could be done by for-profit companies. There is no plan to share with you any revenue generated from products developed using your blood samples.

During this study, if the researchers learn new information that may be important to your general health or to your disease or condition, they will share that information with you.

# Will my information and/or tissue samples ever be used for future research?

In addition, be aware that by agreeing to participate in this study, your information, tissue, leukapheresis product, or blood samples could be used for future research studies or sent to other investigators for future research studies without additional consent from you. These future research studies will be reviewed by an oversight group known as an institutional review board if required by law. The information that identifies you will first be removed from your information or tissue samples. If you do not want your information or tissue samples to be used for future research studies without your consent, you should not participate in this study.

Your anonymized study data and anonymized study samples may be shared with research collaborators which may involve data being transferred outside the US and to commercial partners for the purposes of research.

# Your rights

- You do not have to join this study. You are free to say "yes" or "no".
- If you get sick or hurt in this study, you do not lose any of your legal rights to seek payment by signing this form.

- During the study, we might learn new information that you need to know. For example, some information may affect your health or well-being. Other information might make you change your mind about being in this study. If we learn these kinds of information, we would tell you.
- If you join this study, you would not have to stay in it. You could stop at any time (even before you start). Your regular medical care would not change. You would have no penalty for stopping, but it would be better not to join the study if you think that you would change your mind later.

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Your responsibilities

If you join this study, you would have some responsibilities.

- Follow the schedule of study visits and procedures.
- Takes study medications as directed.
- Prevent pregnancy.
- Tell us about side effects.

#### For more information

If you have questions or concerns about this study, you could talk to your doctor anytime. Other people you could talk to are listed below.

| If you have questions about: | Call: |
|---|---|
| This study (including complaints and requests for information) | 206-667-6909 (Alexandre Hirayama MD; study PI) |
| If you get sick or hurt in this study | 206-606-6000 (IMTX clinic) |
| Your rights as a research participant | 206-667-5900 or email irodirector@fredhutch.org (Director of Institutional Review Office, Fred Hutchinson Cancer Center) |
| Your bills and health insurance coverage | 206-606-6226 (Patient Financial Services) |

Emergency number (24 hours): 206-598-8902

## We would like you to donate some of your tissue samples for other future research

During the study, samples of blood, tumor tissue, leukapheresis product and possible other tissue may be collected from you. We refer to these materials as "samples." After we do tests on your samples in this study, some samples may be left over. We would like you to donate these leftover samples for future research. This may include genetic research.

You do not have to donate your tissue for research. You are free to say yes or no. Your regular medical care will not change. If we want to use your tissue for other research or share it with other scientists for research, an ethics review committee (IRB) will review the request. The IRB will decide if we need to ask for your consent to do the research.

Your donated tissue will be stored in a secure location and will be used for research and for other studies that might help to develop new treatments. These future research and drug development studies may be done by us at Fred Hutch or by for-profit companies including Nektar Therapeutics which funded this study, and its collaborators. Researchers will not report their results to you or your doctor. The research results will not appear in your health record. They will not affect your care.

Research on your tissue may help develop new products. If these products make money, there is no plan to share the money with you.

If you donate your tissue for research, you can change your mind anytime. Just call Dr. Alexandre Hirayama at 206-667-6909 and tell us you do not want us to use your tissue. There is no penalty for changing your mind. Your regular medical care will not change. However, if you do change your mind, we cannot return donated tissue. We may be able to destroy tissue we know is yours. But if it is stored or shared anonymously (without any label saying who it belongs to), we cannot destroy it. In this case it would still be used for research, but no one would know it was yours.

Read each question and think about your choice. When you decide on each question, please circle YES or NO.

| NO. | | | | |
|---|---|---|---|---|
| Do you agree to donate your samples to study cancer and related diseases? Circle and initial one. | | | | |
| YES | NO | Initials: | Date: | |
| Do you agree to donate your samples to study other health problems, such as diabetes, Alzheimer's disease, or heart disease? Circle and initial one | | | | |
| YES | NO | Initials: | Date: | |
| | | | Date: | r research? Circle and |

# **Optional tumor biopsies**

During this study we would like to ask your permission to collect additional tumor biopsies. If you agree to participate, up to 4 additional tumor biopsies will be completed if safe to do so. Biopsies would be done: 1) during pretreatment prior to receiving your chemotherapy and liso-cel infusion; 2) within 4 weeks after you receive your liso-cel infusion 3) within 4 weeks after your first NKTR-255 infusion; and 4) in the event of persistent mass, or your disease relapses or progresses. If at any of these time points you are having a tumor biopsy completed for clinical reasons, we would obtain a sample of that biopsy. You would not have a research biopsy completed in addition. There may be variations in this schedule and your study doctor will discuss with you when this tumor tissue collection procedure may take place.

You do not have to agree to take part in these additional tumor biopsies in order for you to take part in the main study. Your decision to take part is voluntary. If you agree to participate in these optional biopsies you can change your mind at any time and withdraw your permission by letting the study doctor know.

Read the statements below and initial next to the one that applies to you:



# **Signatures**

Please sign below if you:

- have read this form (or had it read to you);
- had the opportunity to ask any questions you have;
- had the opportunity to discuss the research with the person obtaining consent; and
- agree to participate in this study.

| Participant: | | |
|---|---|---|
| Printed Name | Signature | Date |
| <ul><li>have read this fo</li><li>had the opportur</li><li>had the opportur</li></ul> | • • | |
| Printed Name | Signature | Date |
| Relation to the participant | | |
| indicate (1) you were p | resent at the consent discussion consent form, and (3) the participation | ead this written consent form, sign below t<br>in person, (2) you witnessed the verba<br>ant had the opportunity to ask questions an |
| Impartial Witness: | | |
| Printed Name | Signature | <u>Date</u> |

# Researcher's statement

I have discussed the research study, including procedures and risks, with the person signing above. A copy of the signed consent form will be given to the participant.

| Person obtaining consent signature: | | |
|-------------------------------------|-----------|------|
| Printed Name | Signature | Date |

IR file: 10802

Protocol: RG1122036

Current version date: 09/23/2024 Previous version date: 10/24/2023

Copies to: Medical Records, Research File, Participant